CLINICAL TRIAL: NCT02885961
Title: Investigating the Role of the Coagulation Cascade in Idiopathic Pulmonary Fibrosis
Brief Title: The Coagulation Cascade in Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRAS191454
Record Dates: First submitted 2016-08-15; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Idiopathic Pulmonary Fibrosis; IPF; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dabigatran (Other): All patients will be entered into the arm, i.e. this is a single arm study. All patients will complete 2 FDG PET scans. All patients will receive dabigatran (direct thrombin inhibitor) at a dose of 110mg twice daily (oral).
  The drug will be given for 24 days (+/-3 days). The variation in duration reflects that scans are completed Monday to Friday only.
  Interventions: Drug: Dabigatran; Radiation: FDG PET scan

INTERVENTIONS:
Drug: Dabigatran — Anti-coagulant
Radiation: FDG PET scan — Scan using PET combined with a high resolution CT scan (HRCT)

SUMMARY:
The pathogenesis of idiopathic pulmonary fibrosis (IPF) is incompletely understood but recurrent epithelial injury occurs which evokes the coagulation cascade. Thrombin is produced as a result and is over expressed in IPF patients, so may be important in propagating disease activity. We aim to recruit patients with IPF and then complete FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET (positron emission tomography) scans pre and post manipulation of the coagulation cascade to assess the role of this biological pathway in disease activity. Previous studies from our institution have demonstrated increased FDG avidity in the lungs of patients with IPF (assessed using FDG PET scans) but to date the cells and pathways responsible for this signal have not been identified and thus need further exploration.

DETAILED DESCRIPTION:
Patients with IPF who meet all the inclusion criteria (and none of the exclusion criteria) will be assessed and invite to participate.

They will undergo baseline assessment with lung function, 6 minute walk test and health quality assessments.

Blood tests will assess the pro-coagulant state of these individuals. They will undergo a baseline FDG PET scan followed by manipulation of the coagulation cascade with 24 days (+/- 3 days) dabigatran. They will then complete a second FDG PET, health quality assessments and blood tests to demonstrate target engagement.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of IPF based on multi disciplinary meeting discussion following review of the clinical history, characteristic features on HRCT (high resolution CT scan) and/or usual interstitial pneumonia (UIP) histology.
* Written informed consent obtained from subject.

Exclusion Criteria:

* Age <40 or >80 years
* Renal impairment as defined by a creatinine clearance of <30 millilitres/min
* Significant liver impairment with evidence of synthetic dysfunction
* Any contraindication to anti-coagulation including previous life threatening or serious bleed or bleeding tendency.
* Co-administration of any concomitant medications prohibited in full protocol. N-acetyl cysteine, prednisolone up to 10mg daily and pirfenidone are permitted.
* Pregnant, breast feeding or unwilling to practice birth control during participation in the study (females of child bearing age).
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient of the quality of the data.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Demonstrate a change in FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) avidity | Approximately 4 weeks
  FDG avidity describes the degree of tissue uptake of the labelled glucose. It is a numerical continuous variable. It is calculated from the scan using several methods, manually on a workstation and using a mathematical modelling computer programme. The main number generated is called the standardised uptake value (SUV) and the higher the number the higher the metabolic activity in the area. The degree of activity will be quantified for each individual and compared with standard measures of disease activity i.e. lung function measures and quality of life questionnaires. For each individual the change in the SUV measure will be analysed from the scan performed before and then after manipulation of the coagulation cascade.

SECONDARY OUTCOMES:
Demonstrate changes in various coagulation factors | Approximately 4 weeks
  This patient group have demonstrated a hyper coagulable state in a number of previous studies. We will demonstrate this using blood tests prior to administration of dabigatran. The coagulation markers (a blood test, many used in standard clinical practice) will be repeated during treatment to demonstrate target engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna C Porter, PhD FRCP, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No